CLINICAL TRIAL: NCT07348068
Title: The Effect of the Emotional Freedom Technique Applied to Postmenopausal Women Before Probe Curettage on Pain, Anxiety and Vital Signs.
Acronym: EFT-ANXIETY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Elif Elmas, graduate student, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSU-MED-TRIAL-01; 2024/109 (Other: Ethics Committee Protocol Number)
Record Dates: First submitted 2025-01-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: The Effect of Emotional Freedom Technique on Anxiety, Pain, and Vital Signs
Keywords: Anxiety, Pain, and Vital Signs
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: "This study uses a behavioral intervention model in which Emotional Freedom Techniques (EFT) are applied to postmenopausal women prior to a probe curettage procedure to examine its effects on pain, anxiety, and quality of life. EFT is a technique that involves gently tapping on specific acupuncture points while focusing on emotional distress. The intervention aims to reduce anxiety related to pain and improve overall quality of life. The study will evaluate the effectiveness of EFT applied prior to the probe curettage procedure on pain, anxiety, and quality of life during the procedure in postmenopausal women."
Masking Description: "Participants were blinded to the specific details of the procedure being applied, including whether or not the emotional freedom technique (EFT) was used during the probe curettage procedure."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT İNVERTİON GROUP (Experimental): During the initial consultation, the Personal Information Form, SUE Scale, State Anxiety Scale (SAS), Visual Analog Scale (VAS), vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) Monitoring Form will be administered. EFT, which lasts approximately 30-40 minutes, will be administered to women by the researcher. Second measurement: Immediately after EFT, the SUE Scale, State Anxiety Scale (SAS), Visual Analog Scale (VAS), and vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) will be administered again. Following the second measurement, the probe curettage will be performed. Third measurement: During the procedure, the VAS and vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) Monitoring Form will be administered. Fourth measurement: After the probe curettage, women will be given 2 minutes to rest. The Visual Analog Scale (VAS) and vital signs (blood pressure, heart rate, and peripheral oxygen satur
  Interventions: Behavioral: emotional freedom technique
- control group (No Intervention): During the initial consultation, the Personal Information Form, SUE Scale, State Anxiety Scale (SAS), Visual Analog Scale (VAS), vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) Monitoring Form will be administered. Second measurement: The SUE Scale, State Anxiety Scale (SAS), Visual Analog Scale (VAS), and vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) will be administered again simultaneously with the EFT group. Following the second measurement, a probe curettage will be performed. Third measurement: During the procedure, the VAS and vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) Monitoring Form will be applied. Fourth measurement: After the probe curettage, women will be given 2 minutes to rest. The Visual Analog Scale (VAS) and vital signs (blood pressure, heart rate, and peripheral oxygen saturation/SpO2) Monitoring Form will be applied.

INTERVENTIONS:
Behavioral: emotional freedom technique — In this study, the effect of emotional freedom technique on pain, anxiety, and vital signs prior to the probe curettage procedure will be examined. The EFT session will be administered by an EFT specialist approximately 40 minutes prior to the probe curettage procedure by tapping on the tapping points.
  Arms: EFT İNVERTİON GROUP

SUMMARY:
The aim of the study is to examine the effect of the emotional freedom technique applied to postmenopausal women before the probe curettage procedure on pain, anxiety and vital signs.

DETAILED DESCRIPTION:
In this experimentally designed study, it was aimed to examine the effect of the emotional freedom technique applied to postmenopausal women before the probe curettage procedure on pain, anxiety and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Those who are in menopause
* Do not have conditions such as infection, wound or scar in the tapping areas,
* Having no problem communicating in Turkish,
* Those who have not used any analgesic medication in the last 24 hours,
* Those who have not had probe curettage before,
* Volunteer to participate in the study,
* Not using any medication that directly affects vital signs,
* Does not have a disease that would cause problems in feeling pain,
* Not using antidepressants, anxiolytics and sedative agents.

Exclusion Criteria:

* • Those who are not in menopause

  * Women who have had probe curettage before
  * Their general condition deteriorates during the procedure or a different intervention is made with anesthesia,
  * Any complications developed during the procedure,
  * Those who experienced syncope during the procedure and the procedure was continued with general/local anesthesia,
  * Having a psychiatric problem,
  * Analgesic medication used during the procedure,
  * Having cognitive, affective, perceptual problems.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 132 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline (pre-procedure) and during the probe curettage procedure.
  Pain intensity will be assessed using the Visual Analogue Scale (VAS), a numeric rating scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory - State Version (STAI-I) | Baseline (pre-procedure) and immediately post-procedure.
  Anxiety levels will be assessed using the State-Trait Anxiety Inventory - State Version (STAI-I), which measures situational anxiety at a specific point in time. The scale consists of 20 items, with total scores ranging from 20 to 80. Higher scores indicate greater levels of anxiety.
Systolic and Diastolic Blood Pressure | Baseline (pre-procedure), during the probe curettage procedure, and immediately post-procedure (within 2 minutes after completion).
  Systolic and diastolic blood pressure will be measured to evaluate physiological responses associated with the probe curettage procedure and the effect of the Emotional Freedom Technique (EFT).
Heart Rate | Baseline (pre-procedure), during the probe curettage procedure, and immediately post-procedure (within 2 minutes after completion).
  Heart rate will be measured to assess autonomic physiological responses related to anxiety, pain, and procedural stress during the probe curettage procedure.
Peripheral Oxygen Saturation (SpO₂) | Baseline (pre-procedure), during the probe curettage procedure, and immediately post-procedure (within 2 minutes after completion).
  Peripheral oxygen saturation will be measured to monitor respiratory and physiological stability during and after the probe curettage procedure.

OTHER OUTCOMES:
State-Uncertainty Emotion (SUE) Scale | Baseline (pre-procedure) and immediately post-procedure (within 2 minutes after completion).
  Emotional distress related to uncertainty will be assessed using the State-Uncertainty Emotion (SUE) Scale. The scale is scored on a numeric scale from 0 to 10, where higher scores indicate greater emotional distress and uncertainty.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - kahramanmaraş NFK Obstetrics and Pediatrics Hospital Additional Service Building, Kahramanmaraş, Kahramanmaraş
  - Kahramanmaraş Sütçü Imam Üniversitesi, Kahramanmaraş, Kahramanmaraş
  - Kahramanmaraş Sütçü Imam Üniversitesi, Kahramanmaraş

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to privacy concerns and to ensure confidentiality of personal information. Additionally, the data is collected for a specific study and will not be made available for secondary analyses.

REFERENCES:
- See also: "This link redirects to the website of Sütçü İmam University." — https://www.ksu.edu.tr/